CLINICAL TRIAL: NCT06505902
Title: Pulmonary Diffusing Capacity During Incremental Exercise in COPD: A Case-Control Study
Brief Title: Pulmonary Diffusing Capacity During Incremental Exercise in COPD
Acronym: DiffLung3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Milan Mohammad, Medical Doctor, Principal Investigator, PhD-student at the Department of Physical Activity Research center, Copenhagen, Denmark., Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-24025935
Record Dates: First submitted 2024-07-08; First posted 2024-07-17 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: COPD; Healthy; Lung Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Matched case-control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COPD-patients (Experimental): COPD-patients during diffusing capacity measurement during incremental exercise
  Interventions: Other: Exercise
- Matched healthy volunteers (Experimental): Healthy matched controls during diffusing capacity measurement during incremental exercise
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise by bicycle and performing diffusing capacity measurements at the same time with arterial blood gasses.

SUMMARY:
Background:

The combined measurement of pulmonary diffusing capacity for carbon monoxide (CO) and nitric oxide (NO) (DL,CO,NO) has recently been standardized and validated for clinical use. It involves a noticeably short breath-hold time (≤5 seconds), making it feasible to perform on patients with chronic obstructive pulmonary disease (COPD). These patients have lower diffusing capacity and are unable to increase it during exercise, which is thought to be caused by changes in pulmonary perfusion potentially leading to exertional dyspnea. The aim of the present study is to examine whether pulmonary diffusing capacity for incremental exercise differs between patients with COPD and matched healthy controls.

Methods:

Inclusion of 12 individuals with mild-to-severe COPD and 12 healthy age- and sex-matched controls.

Design: Case-control study

Intervention: DL,CO,NO and arterial blood gases will be measured during exercise at a bicycle ergometer at 0, 20, 40, 60 and 80% of the individual's maximal workload.

Sample size: To detect a 15 mmol min-1 kPa-1 difference in DL,NO between groups at 60% of maximal workload, with a power of 90% and a significance level of 0.05, at least 12 subjects are required in each group. To account for potential dropouts, power will be permitted to decrease to 80%, corresponding to a total of 10 subjects in each group.

Statistical design: Linear mixed effect model and pairwise testing of estimated marginal means.

Perspective: This study will add to the understanding exertional dyspnoea in patients with COPD.

DETAILED DESCRIPTION:
Introduction and background A pattern that applies to the majority of the more than 250 million people who suffer from chronic obstructive pulmonary disease (COPD) worldwide, is a downward spiral of exertional dyspnoea to poor quality of life, invalidity, and early death. A critical mechanism of exertional dyspnoea in these patients is thought to be reduced alveolar-capillary reserve, that is, a reduced ability to recruit and distend the pulmonary capillary bed to increase diffusing capacity upon an increase in cardiac output, which may be assessed by measuring the dual test pulmonary diffusing capacity (DL,CO,NO) during exercise. This technique permits up to 12 repeated manoeuvres within a session without affecting measurements, and it is thus ideal for assessing acute changes in pulmonary diffusing capacity and its components during various physiological manoeuvres. With this technique, the investigators have recently documented that alveolar-capillary recruitment, assessed by the change in the pulmonary diffusing capacity for nitric oxide (DL,NO) at a fixed workload of 60% of maximum, is blunted in COPD, seemingly in a severity-dependent fashion (unpublished observations). However, it is unknown whether this is already evident at low workloads, and/or whether it persists at near-maximal workloads, and it remains to be established to which extent this has an impact on pulmonary gas exchange, conventionally measured by the alveolar-arterial oxygen difference.

Aim The overall aim is to determine whether and how alveolar-capillary recruitment during incremental exercise differs between patients with mild-to-moderate COPD and healthy individuals.

Study design and recruitment 12 patients with mild-to-moderate COPD and 12 healthy age- and sex-matched controls will be included in the study, where DL,CO,NO will be measured at rest and during incremental workloads. Visit 0 consist of medical health interview and brief examination including blood pressure, heart rate and ECG measurement to investigate inclusion and exclusion criteria. Baseline measurements (Visit 1) will be performed to assess fitness and cardiopulmonary health status for the included patients and participants. The baseline measurements include cardiopulmonary exercise testing, lung function testing (dynamic spirometry, whole-body plethysmography and 10-second single-breath diffusing capacity for carbon monoxide), and an assessment of body composition. On Visit 2, which is at least two days later, an arterial catheter is inserted, after which DL,CO,NO and arterial blood gases are measured at rest, and at 20, 40, 60, and 80% of maximal workload on a bicycle ergometer, as determined during the cardiopulmonary exercise text on Visit 1.

Sample size Based on unpublished data in which a difference in DL,NO (mmol min-1 kPa-1) between COPD and control at 60% of maximal workload during cycling exercise, the power calculation was based on a two-sided independent samples t-test, with a power of 90% and a significance level (alpha) of 0.05. To detect a 15 mmol min-1 kPa-1 difference in DL,NO between groups at 60% of maximal workload, with a power of 90% and a significance level of 0.05, at least 12 subjects are required in each group. To account for potential dropouts, power will be permitted to decrease to 80%, corresponding to a total of 10 subjects in each group.

Statistical procedure The investigators will perform a linear mixed effect model with group and time as factors with participant as random effect accounting for repeated measures. The investigators will then perform pairwise testing of estimated marginal means from our mixed effect model to test for between group differences and within group differences. The investigators will perform Holm correction due to multiple testing.

General information This study is novel as it investigates pulmonary capillary recruitment in COPD, which is thought to be an important mechanism of exertional dyspnoea, which have primarily only been discussed in theoretical terms in previous studies. This study will be conducted in accordance with the regional ethical committee and the Declaration of Helsinki. Informed consent will be obtained from all study participants before enrolment and baseline testing.

Significance, novelty and expected impact The physiological assessments that are evaluated in the present study have the potential to be used provide information on the cause of dyspnoea in the individual COPD patient. This is relevant for the understanding of basic respiratory physiology and for designing future studies with interventions that aim to affect pulmonary capillary recruitment in COPD.

ELIGIBILITY:
Inclusion criteria for COPD patients

* Men and women
* 40-80 years
* Mild to severe COPD (GOLD stage I to IIII)

Inclusion criteria for healthy participants

* Men and women
* Age +/- 3 years of an included COPD patient

Exclusion criteria for COPD patients

* Known ischaemic heart disease
* Known heart failure
* Cardiac arrythmias
* Dementia or other severe neurological disease
* Known vascular ischaemic disease
* Symptoms of infection (bacterial/viral) within 2 weeks prior to the study
* Pregnancy

Exclusion criteria for heathy controls

* COPD
* Known ischaemic heart disease
* Known heart failure
* Cardiac arrythmias
* Dementia or other severe neurological disease
* Known vascular ischaemic disease
* Symptoms of infection (bacterial/viral) within 2 weeks prior to the study
* Pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome | Measured at day 2
  Between-group difference in the change in DL,NO from rest to exercise as a function of workload

SECONDARY OUTCOMES:
Key secondary outcome | Measured at day 2
  Between-group difference in the change of the alveolar-arterial oxygen difference from rest to exercise as a function of workload
Other secondary outcome | Measured at day 2
  Between-group difference in the change in DL,NO from rest to exercise as a function of VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change of the alveolar-arterial oxygen difference from rest to exercise as a function of VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in cardiac output from rest to exercise as a function of workload
Other secondary outcome | Measured at day 2
  Between-group difference in the change in stroke volume from rest to exercise as a function of workload
Other secondary outcome | Measured at day 2
  Between-group difference in the change in heart rate from rest to exercise as a function of workload
Other secondary outcome | Measured at day 2
  Between-group difference in the change in mean arterial blood pressure from rest to exercise as a function of workload
Other secondary outcome | Measured at day 2
  Between-group difference in the change in cardiac output from rest to exercise as a function of VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in stroke volume from rest to exercise as a function of VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in heart rate from rest to exercise as a function of VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in mean arterial blood pressure from rest to exercise as a function of VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in PaO2 from rest to exercise as a function of workload and VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in SaO2 from rest to exercise as a function of workload and VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in PaCO2 from rest to exercise as a function of workload and VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in pH from rest to exercise as a function of workload and VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in base excess from rest to exercise as a function of workload and VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in lactate from rest to exercise as a function of workload and VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in respiratory rate from rest to exercise as a function of workload and VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in DL,CO,5s from rest to exercise as a function of workload and VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in DM from rest to exercise as a function of workload and VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in VC from rest to exercise as a function of workload and VO2
Other secondary outcome | Measured at day 2
  Between-group difference in the change in VA from rest to exercise as a function of workload and VO2

OTHER OUTCOMES:
Exploratory outcomes | Measured at day 2
  Between-group difference in time constant (phase 2) (s) from VO2kinetics
Exploratory outcomes | Measured at day 2
  Between-group difference in mean response time (s) from VO2kinetics
Exploratory outcomes | Measured at day 2
  Between-group difference in amplitude (mLO2/min) from VO2kinetics
Exploratory outcomes | Measured at day 2
  Between-group difference in steady state gain (mLO2•min-1•watt-1) from VO2kinetics
Exploratory outcomes | Measured at day 2
  Between-group difference in time delay (phase 1) (s) from VO2kinetics
Exploratory outcomes | Measured at day 2
  Between-group difference in relative (mL/kg/min) VO2peak
Exploratory outcomes | Measured at day 2
  Between-group difference in absolute (mL/min) VO2peak
Exploratory outcomes | Measured at day 2
  Between-group difference in ventilatory threshold (%)
Exploratory outcomes | Measured at day 2
  Between-group difference in ventilatory reserve (%)
Exploratory outcomes | Measured at day 2
  Between-group difference in resistance (Rrs, R5-R20) measured by IOS
Exploratory outcomes | Measured at day 2
  Between-group difference in reactance (Xrs, X5) measured by IOS
Exploratory outcomes | Measured at day 2
  Between group difference in mean arterial pressure (MAP) as a function of workload.
Exploratory outcomes | Measured at day 2
  Between group difference in systolic blood pressure (SBP) as a function of workload.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Mohammad, MD, Principal Investigator — Centre for Physical Activity Research, Rigshospitalet
Locations (1):
- Center for Aktiv Sundhed (CFAS), Rigshospitalet, Copenhagen, Denmark., Copenhagen, København Ø, Denmark